CLINICAL TRIAL: NCT03325348
Title: Oral Nifedipine Versus IV Labetalol in Treatment of Severe Pre Eclampsia in Pregnancy
Brief Title: Oral Nifedipine Versus IV Labetalol in Severe Pre Eclampsia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, Tayyiba Wasim, professor obs Gynecology, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB/2017/306/SIMS
Record Dates: First submitted 2017-09-30; First posted 2017-10-30 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Severe Pre-Eclampsia, Antepartum
Keywords: Severe Pre eclampsia; Nifidepine; Labetalol
MeSH Terms: conditions — Pre-Eclampsia | interventions — Nifedipine; Labetalol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Nifedipine (Experimental): Nifedipine 10mg oral tablet & 1ml 0.9%N/Saline will be given every 15 minutes up till one hour
  Interventions: Drug: Nifedipine 10 mg
- IV Labetalol (Active Comparator): IV labetalol 20 mg and mint tablet will be given every 15 minutes up till one hour
  Interventions: Drug: Labetalol

INTERVENTIONS:
Drug: Nifedipine 10 mg — Nifedipine 10mg oral tablet with 1 ml 0.9% n/saline will be given to patients every 15 min uptil one hour
  Other Names: Cap nefidil 10 mg
  Arms: Oral Nifedipine
Drug: Labetalol — IV labetalol 20 mg & mint tablet will be given to patients every 15 min until one hour
  Other Names: Labetalol Hydrochloride injection
  Arms: IV Labetalol

SUMMARY:
OBJECTIVE: To determine the efficacy of nifedipine and labetalol in terms of control of BP in pre eclamptic pregnant patients

Design: Randomised control trial

SETTING: Department Obstetrics & gynaecology, Services Hospital, Services Institute of Medical Sciences. Lahore

POPULATION: Pregnant patients with BP 160/110 or symptoms of severe preeclampsia

METHODS: Patients are randomised to receive nifedipine (10 mg tablet, orally, up to five doses) and intravenous placebo saline injection or intravenous labetalol injection (in an escalating dose regimen of 20, 40, 80, 80 and 80 mg) and a placebo tablet every 15 minutes until the target blood pressure of ≤140/90mmHg is achieved. Crossover treatment is given if the initial treatment regimen is unsuccessful

DETAILED DESCRIPTION:
Gestational hypertension is associated with increased risk of maternal morbidity and mortality. Parenteral therapy needs more resources, more monitoring and supervision. Oral therapy is cheap, easily available, easy to administer especially in resource constrained settings

OBJECTIVE: To determine the efficacy of nifedipine and labetalol in terms of control of BP in pre eclamptic pregnant patients

Design: Randomised control trial SETTING: Department Obstetrics & gynaecology, Services Hospital, Services Institute of Medical Sciences.Lahore POPULATION: Pregnant patients with BP 160/110 mm Hg or symptoms of severe preeclampsia

METHODS: Patients are randomised to receive nifedipine (10 mg tablet, orally, up to five doses) and intravenous placebo saline injection or intravenous labetalol injection (in an escalating dose regimen of 20, 40, 80, 80 and 80 mg) and a placebo tablet every 15 minutes until the target blood pressure of ≤140/90mmHg is achieved. Crossover treatment is given if the initial treatment regimen is unsuccessful

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24 to 41 weeks
* BP > 160/110 mm Hg with proteinuria
* Patients with S/S of imminent eclampsia as headache, visual disturbance.

Exclusion Criteria:

* Gestational age < 24 wks
* Non proteinuric chronic hypertension
* Eclampsia
* Cardiac patients, asthma, severe renal disease, allergy to Nifedipine or Labetalol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 194 (Estimated)
Dates: Start 2017-02-23 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-01-15 (Estimated)

PRIMARY OUTCOMES:
Time taken for Blood Pressure control | 60 minutes
  Time taken to control Blood pressure will be measured

SECONDARY OUTCOMES:
Fetal distress | Labour
  Fetal distress will be measured by abnormalities of fetal heart rate of fetus or passage of meconium.
  of Meconium
Neonatal Intensive Care Unit admission, | From Birth till 7 days
  If neonate needs Neonatal Intensive Care Unit admission for more than 12 hours
perinatal death | From birth to 7 days
  If death of baby occurs in utero or within 7 days of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan